CLINICAL TRIAL: NCT01695707
Title: Assessing the Impact of Pioglitazone on Skin Barrier Function in Atopic Dermatitis Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient Funding.
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Lisa Beck, Professor of Dermatology, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RSRB00041078; 1R21AR062357 (NIH)
Record Dates: First submitted 2012-09-26; First posted 2012-09-28 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Atopic Dermatitis
Keywords: atopic dermatitis; eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Subjects randomized to placebo will receive opaque size "00" gelatin capsules containing 240mg lactose. As with the intervention group, 1 capsule will be taken by each day throughout the treatment period.
  Interventions: Drug: Placebo (for pioglitazone)
- Pioglitazone (Experimental): Subjects randomized to pioglitazone will receive opaque size "00" gelatin capsules containing pioglitazone. For the first 3 weeks, capsules will contain 30 mg pioglitazone. For the remaining 9 weeks of the treatment period, capsules will contain 45 mg pioglitazone unless subjects are unable to tolerate this increased dose.
  One capsule will be taken by each day throughout the treatment period.
  Interventions: Drug: Pioglitazone

INTERVENTIONS:
Drug: Pioglitazone — see Arm Description
  Other Names: Actos
  Arms: Pioglitazone
Drug: Placebo (for pioglitazone) — see Arm Description
  Arms: Placebo

SUMMARY:
Many patients with eczema (atopic dermatitis) have an inherent defect in their skin barrier as demonstrated by high water loss. In laboratory conditions, studies have shown that pioglitazone restores the skin barrier function in skin from eczema patients. The purpose of this study is to determine if taking pioglitazone improves the skin barrier function in people with eczema.

DETAILED DESCRIPTION:
Enrolled patients will be randomized to either placebo or pioglitazone. Each randomized subject will have a skin biopsy and skin irritancy assay performed prior to treatment and at the end of 12 weeks of treatment. Noninvasive barrier measurements including transepidermal water loss will be recorded at all study visits.

ELIGIBILITY:
Inclusion Criteria:

* i. Moderate to Severe AD: EASI ≥ 10 ii. Active Atopic Dermatitis: Subjects must have within the last 3 months according to medical records or by medical exam of the investigator:

  * Pruritus
  * Eczema (acute, subacute, chronic)

I. Typical morphology and age-specific patterns - Patterns include (1) facial, neck, and extensor involvement in infants and children, (2) current or prior flexural lesions in any age group, (3) sparing groin and axillary regions.

II. Chronic or relapsing history

iii. Extrinsic they must also meet both of the following: serum total IgE ≥ 1.5 S.D. greater than the age-matched norms and positive multi-allergen RAST (Phadiatop).

Additionally, subjects must have TEWL of nonlesional skin of upper arm that is ≥ 8 gm/m2/h at screening visit. This is to ensure that we are in fact studying the subset of AD subjects who have a skin barrier defect.

Exclusion Criteria:

* Unwillingness or inability to complete the Informed Consent process
* Subjects with a history of keloid formation
* History of lidocaine or Novocain allergy
* Subjects with a systemic infection requiring a course of systemic antibiotics or antivirals within the last 2 weeks
* Subjects with MD diagnosed Type 1 or 2 diabetes mellitus
* Subjects with NYHA class III or IV cardiac status
* Subjects with a history of liver disease (EtOH, viral hepatitis, drug-induced hepatitis or other)
* Subjects with evidence of an underlying systemic disease based on history and physical (other than the above diagnostic categories (and associated allergic disorders), or well-controlled hypertension, or hyperlipidemia).
* History of cancer other than nonmelanomatous skin cancer or cervical dysplasia
* Participants enrolled while on a systemic treatment for their atopic dermatitis (e.g. cyclosporine, mycophenolate mofetil) must remain on a stable dose for the duration of the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-03; Primary Completion 2014-01 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Noninvasive barrier measurements (TEWL)
  Transepidermal Water Loss (TEWL) will be measured at multiple time points throughout the study as a surrogate for skin barrier integrity.
Transepithelial electrical resistance (TEER) and permeability
  Skin biopsies will be performed twice during the study. The integrity of the skin barrier will be assessed in the lab by transepithelial electrical resistance (TEER) and permeability of the biopsy specimens.
mRNA
  Ex vivo assessment of mRNA expression of key epidermal barrier proteins will also be performed on the biopsy specimens.

SECONDARY OUTCOMES:
Skin Irritancy
  The clinical efficacy of PIO will be assessed by quantifying the skin response to a model irritant, sodium lauryl sulphate (SLS) at several time points. Subjects will be exposed for 24 h on the dominant inner arm to SLS at three concentrations (wt/vol in water - 0.125, 0.5 and 2%) (Fluka) using standard patch test reagents (Finn chambers of 18-mm diam, Filter Discs & Scanpor tape). Before application and at several time points after removal, TEWL and erythema will be measured at the exposed site and at a control site. Erythema will be measured using a colorimeter (Minolta CR-200).

CONTACTS AND LOCATIONS:
Overall Officials: Lisa A Beck, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States